CLINICAL TRIAL: NCT00966212
Title: Reducing Alcohol & Risks Among Young Females
Brief Title: Parent Education for Young Teen Females
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Education Development Center, Inc. (Industry)
Responsible Party: Principal Investigator, Lydia O'Donnell, Senior Scientist, Education Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6241; 1R01AA014515 (NIH)
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- health promotion materials (No Intervention)
- print parent education (Active Comparator)
  Interventions: Behavioral: parent education

INTERVENTIONS:
Behavioral: parent education — Especially for Daughters audio-cd parent education
  Arms: print parent education

SUMMARY:
The study has the potential to improve understanding of the link between early alcohol and sexual initiation and to provide a proven, selective, female-focused intervention for addressing these risks. The goal is to set young women on a course that protects their health and reduces the burden that problem drinking and HIV disease is taking on African American and Latino communities.

DETAILED DESCRIPTION:
The aims of this study are to to characterize and address the combined risks of early alcohol use and early sexual initiation within a population of urban African American and Latina adolescent females who are at high risk for HIV, AIDS, and other STI. Past research by the investigative team has documented that nearly 10% of females in our target population have initiated sex by fall of 7th grade and more than half have done so by spring of 10thgrade. Although alcohol use is more comparable with national figures, the combination of early alcohol and early sexual initiation is troubling, yet under-addressed by existing interventions. We will develop and test an intervention that builds upon a promising strategy for influencing adolescents: parent education. Three parenting mechanisms shown to influence adolescent risk behavior are targeted: parental monitoring, household rule setting, and communication. Informed by a community advisory board and a series of focus groups, a set of three audio-cds for parents of young adolescents will be developed. Through dramatic role-model stories, these CDs will help parents address alcohol prevention and the link between early alcohol use and sexual initiation and risk taking. Families and middle school daughters will then be enrolled into a randomized pilot test of the intervention's efficacy. Parent and student surveys will be conducted at baseline and 3-month post-intervention follow up to assess whether the intervention is beneficial in terms of promoting positive parenting practices, positive attitudes toward healthy behaviors, and reducing girls' risks.

ELIGIBILITY:
Inclusion Criteria:

* 8th grade girls and parents at participating schools

Exclusion Criteria:

* Non-English speaking

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
positive parenting practices | 3 months
alcohol use | 3 months
risk behaviors | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Education Development Center, Newton, Massachusetts, United States